CLINICAL TRIAL: NCT04824651
Title: Covid-19 Vaccine Cohort in Specific Populations
Acronym: COV-POPART
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS0001S
Record Dates: First submitted 2021-03-25; First posted 2021-04-01 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Immune Deficiency
Keywords: COVID-19 vaccine; Immunogenicity; Immunosuppression; Population at risk
MeSH Terms: conditions — Immunologic Deficiency Syndromes | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Laboratory tests:
  PCR SARS-Cov2 (Severe Acute Respiratory Syndrome-related Coronavirus-2) Serology (research Anti-Spike - Anti RBD (Receptor Binding Domain) - Anti NCP (Nucleoprotein) + neutralization tests) peripheral blood mononuclear cell : PBMC (immunity testing) total blood for DNA bank Plasma bank RNA bank
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (15):
- Solid cancer: objective : 800 participants for adult cohort, 100 for pediatric cohort (solid cancer and malignant hemopathy)
  Interventions: Biological: COVID-19 vaccine
- Solid organ transplantation: objective : 700 participants for adult cohort, 50 for pediatric cohort
  Interventions: Biological: COVID-19 vaccine
- Allogeneic hematopoietic stem cell transplantation: objective : 350 participants for adult cohort, 50 for pediatric cohort
  Interventions: Biological: COVID-19 vaccine
- Chronic renal failure: Patients with chronic renal failure stage 4, 5 who receive dialysis or not. objective : 350 participants for adult cohort, 30 for pediatric cohort
  Interventions: Biological: COVID-19 vaccine
- Autoimmune and autoinflammatory systemic diseases: Systemic lupus erythematosus ,Systemic Vasculitides,... objective : 750 participants for adult cohort, 130 for pediatric cohort
  Interventions: Biological: COVID-19 vaccine
- Multiple sclerosis/ Neuromyelitis optica diseases: MS defined by Mac Donald et al. 2017 and Neuromyelitis optica defined by Wingerchuk et al. 2015 ; objective : 600 participants for adult cohort
  Interventions: Biological: COVID-19 vaccine
- Chronic inflammatory rheumatism: Ankylosing spondylitis and rheumatoid polyarthritis objective : 600 participants for adult cohort
  Interventions: Biological: COVID-19 vaccine
- Hypogammaglobulinemia: objective : 300 participants for adult cohort
  Interventions: Biological: COVID-19 vaccine
- Obese non diabetic: BMI ≥ 30 objective : 1400 participants for adult cohort, 100 for pediatric cohort
  Interventions: Biological: COVID-19 vaccine
- Diabetic (type I and II) obese or not: objective : 1400 participants for adult cohort, 100 for pediatric cohort
  Interventions: Biological: COVID-19 vaccine
- People living with HIV-1: objective : 1400 participants for adult cohort
  Interventions: Biological: COVID-19 vaccine
- Senior group (free from chronic conditions of interest listed above): ≥75 years objective : 450 participants for adult cohort
  Interventions: Biological: COVID-19 vaccine
- Control group (free from chronic conditions of interest listed above): 18 to 74 years objective : 1400 participants for adult cohort, 100 for pediatric cohort (from 5 to 17 years old)
  Interventions: Biological: COVID-19 vaccine
- Control AZ-PF group (free from chronic conditions of interest listed above): Participants with first dose of Astra-Zeneca vaccine AZD1222 and second dose of Pfizer ARNm vaccine BNT162b2 objective : 200 participants for adult cohort
  Interventions: Biological: COVID-19 vaccine
- Major sickle cell syndrome: 100 for pediatric cohort (from 5 to 17 years old)
  Interventions: Biological: COVID-19 vaccine

INTERVENTIONS:
Biological: COVID-19 vaccine — Vaccination done as part of France's COVID-19 Vaccination Campaign

SUMMARY:
Multicentre national cohort study with prospective data collection and biological specimen collection.

Ancillary study in this cohort : pediatric cohort with participants from 5 to 17 years old.

Enrollment complete for adult cohort. Active recruting for ancillary pediatric cohort.

DETAILED DESCRIPTION:
Primary Objective

1.Evaluate in a standardized manner in each subpopulation the humoral immune response to Covid-19 vaccination at 1, 6, 12, 24 months (M) after the last dose of vaccine (1 or 2 dose schedule depending on the vaccines) and standardized assessment of the humoral response 1 month after receipt of the third injection in participants receiving a third injection as recommended

Secondary objectives

1. Evaluate the cellular immune response to Covid-19 vaccination at Inclusion, 6 and 24 months after the first injection (single-injection scheme) or after the second injection of the vaccine (two or three-injections regimens) in each subpopulation
2. Compare the humoral immune response at 1, 6, 12, 24 months after the first injection (one-injection scheme) or after the second injection of vaccine (two- or three-injections regimens) of each subpopulation with a control group of subjects without the chronic diseases of interest and from any other diseases or treatment taht may have an influence on the immune response.
3. Compare the humoral immune response after 3 injections (1 month after the third dose) to that after 2 injections (1 month after the second dose) in participants with received a third injection as current recommendations
4. In each subpopulation, study the factors associated with the humoral immune response at 1 month and the persistence of the humoral immune response at 6, 12, 24 months as a function of age, stage of disease, treatments, type of vaccine (as well as characteristics specific to the subpopulations studied)
5. Evaluate and characterize the humoral immune response for participants who received a booster dose with mRNA vaccine acording to recommendations in force
6. Compare the humoral immune response between different specific subpopulations
7. Describe the seroconversion for anti-nucleoprotein antibodies
8. Immuno-virologically characterize vaccine failures (SARS-CoV2 infection) during follow-up
9. Identify genetic determinants of the immune response based on the underlying pathology and ongoing treatments if applicable (response and resistance to vaccination)

Specifics secondary objectives for participants with the first dose of Astra-Zeneca vaccine and the second dose of Pfizer vaccine

1. Evaluate the humoral and the cellular immune response to Covid-19 vaccination with this vaccination schedule
2. Evaluate the clinical reaction (local and generale) after this vaccination schedule

ELIGIBILITY:
These eligibility criteria only concern the adult cohort.

INCLUSION CRITERIA :

General inclusion criteria for all patients of all groups

* Be 18 years or older
* Get vaccinated against Covid-19 as part of the national vaccination campaign or having already received a first or second vaccine injection as part of the national vaccination campaign
* Accept the conditions of participation corresponding to each sub-population
* Commit to respecting the schedule of visits provided in the research protocol
* Plan to reside in France for at least 2.5 years from inclusion date
* Give their free, informed and written consent (at the latest on the day of inclusion and before any examination / samples) by signing the consent form
* Be a member of or beneficiary of a social security scheme (State Medical Aid is not a social security scheme).

General inclusion criteria for patients with a chronic condition of interest

* Present at least one pathology listed
* If the participant is participating in the in-depth immunology and virology study, they must have only one of the pathology of interest listed

Inclusion criteria for control subjects • Be free from the chronic conditions of interest listed or other chronic conditions/treatment that may affect the immune response

Inclusion criteria for control subjects free from chronic conditions of interest and with first injection with Astra-Zeneca vaccine AZD1222 and second injection with Pfizer ARNm vaccine BNT162b2

• Be vaccinated with a first injection with Astra-Zeneca vaccine AZD1222 and a second injection with Pfizer ARNm vaccine BNT162b2

NON INCLUSION CRITERIA :

General non inclusion Criteria for all participants of all groups

* Be under protective supervision (guardian or curatorship)
* Being a pregnant or breastfeeding woman
* Present a contraindication to Covid-19 vaccination : Have a known or suspected allergy to any component of the vaccine, Have had at-risk contact with a confirmed Covid-19 person in the last 7 days, Have presented clinical signs suggestive of Covid-19 in the last 7 days, Have an acute febrile episode on inclusion / vaccination, Have received a vaccine in the last 15 days ...
* Have had a documented Covid-19 Infection (PCR or antigenic test)
* Refuse that their Social Security number is collected for accessing the National Health Data System (NSDS)/Data Health Hub national health databases
* For safety reasons, must agree to not enter in a vaccine clinical trial during the entire period of inclusion and follow-up of the research

Specific non inclusion criteria for PLWHIV

* Being infected with HIV-2
* Presenting another cause for immunosuppression (undergoing immunosuppressive treatment, biotherapy)
* Presenting a non controlled opportunistic infection

Specific non-inclusion criteria for control subjects

* Have one or more of the chronic conditions of interest listed or affected by any other pathology or treatment that may affect the immune response (autoimmune/inflammatory pathology or immune deficiency not listed, liver failure, immunosuppressive therapy (like oral corticosteroids at >= 10 mg/d Prednisone equivalent for more than 15 days) or radiotherapy within 6 months prior to inclusion or planned for the duration of the study)
* Life expectancy of less than 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 6110 participants are inclued in the adult cohort.
  Enrollment objective in the ancillary study (pediatric cohort) from 5 to 17 years old (active enrollment): 810.
  The specific populations of the study for adult cohort:
  Patients with solid cancer solid organ transplant patients Allogeneic hematopoietic stem cell transplant patients Patients with chronic kidney failure disease and dialysis Patients with Multiple Sclerosis / Neuromyelitis optica spectrum disorder Patients with Chronic inflammatory rheumatism Patients with Autoimmune and autoinflammatory systemic diseases Patients with Hypogammaglobulinemia Patients obese non diabetic Patients diabetic (type I and II) obese or not People with HIV-1 (only)
  Control group (free from chronic conditions of interest listed above):
  18 to 74 years
  ≥75 years (senior group) Vaccination schedule with Astra-Zeneca vaccine first dose and Pfizer vaccine second dose
Sampling Method: Non-Probability Sample
Enrollment: 6920 (Estimated)
Dates: Start 2021-03-25 (Actual); Primary Completion 2024-06-25 (Estimated); Study Completion 2024-06-25 (Estimated)

PRIMARY OUTCOMES:
These primary outcome only concern the adult cohort. Humoral immunity to Covid-19 vaccination using 2 serological criteria: | before the second injection (if applicable)
  * Anti-Spike (test 1) and anti RBD (test 2) antibodies (quantitative Elisa)
  * Seroneutralization, by conventional in vitro seroneutralization test, for participants having test 1 and / or test 2 positive: percentage of patients with a neutralizing antibody titre specific to SARS-CoV-2 ≥20.
  Seroneutralization, by neutralization test on SARS-CoV-2 variants, in the first 50 participants included by subpopulation and with test 1 and / or test 2 positive: SARS-CoV-2 specific neutralizing antibodies titre
Humoral immunity to Covid-19 vaccination using 2 serological criteria: | Month 1
  * Anti-Spike (test 1) and anti RBD (test 2) antibodies (quantitative Elisa)
  * Seroneutralization, by conventional in vitro seroneutralization test, for participants having test 1 and / or test 2 positive: percentage of patients with a neutralizing antibody titre specific to SARS-CoV-2 ≥20.
  Seroneutralization, by neutralization test on SARS-CoV-2 variants, in the first 50 participants included by subpopulation and with test 1 and / or test 2 positive: SARS-CoV-2 specific neutralizing antibodies titre
Humoral immunity to Covid-19 vaccination using 2 serological criteria: | Month 1 after the third dose (if applicable)
  * Anti-Spike (test 1) and anti RBD (test 2) antibodies (quantitative Elisa)
  * Seroneutralization for participants having test 1 and / or test 2 positive: percentage of patients with a titre ≥40
  * Titre of neutralizing antibodies for participants having test 1 positive (with conventionnal in vitro neutralization test and neutralization test on variants of SARS-CoV-2)
Humoral immunity to Covid-19 vaccination using 2 serological criteria: | Month 6
  * Anti-Spike (test 1) and anti RBD (test 2) antibodies (quantitative Elisa)
  * Seroneutralization, by conventional in vitro seroneutralization test, for participants having test 1 and / or test 2 positive: percentage of patients with a neutralizing antibody titre specific to SARS-CoV-2 ≥20.
  Seroneutralization, by neutralization test on SARS-CoV-2 variants, in the first 50 participants included by subpopulation and with test 1 and / or test 2 positive: SARS-CoV-2 specific neutralizing antibodies titre
Humoral immunity to Covid-19 vaccination using 2 serological criteria: | Month 12
  * Anti-Spike (test 1) and anti RBD (test 2) antibodies (quantitative Elisa)
  * Seroneutralization, by conventional in vitro seroneutralization test, for participants having test 1 and / or test 2 positive: percentage of patients with a neutralizing antibody titre specific to SARS-CoV-2 ≥20.
  Seroneutralization, by neutralization test on SARS-CoV-2 variants, in the first 50 participants included by subpopulation and with test 1 and / or test 2 positive: SARS-CoV-2 specific neutralizing antibodies titre
Humoral immunity to Covid-19 vaccination using 2 serological criteria: | Month 24
  * Anti-Spike (test 1) and anti RBD (test 2) antibodies (quantitative Elisa)
  * Seroneutralization, by conventional in vitro seroneutralization test, for participants having test 1 and / or test 2 positive: percentage of patients with a neutralizing antibody titre specific to SARS-CoV-2 ≥20.
  Seroneutralization, by neutralization test on SARS-CoV-2 variants, in the first 50 participants included by subpopulation and with test 1 and / or test 2 positive: SARS-CoV-2 specific neutralizing antibodies titre
Percentage of participants seroconverting for Anti Nucleoprotein antibodies | Inclusion
  (qualitative Elisa)
Percentage of participants seroconverting for Anti Nucleoprotein antibodies | before the second injection (if applicable)
  (qualitative Elisa)
Percentage of participants seroconverting for Anti Nucleoprotein antibodies | Month 1
  (qualitative Elisa)
Percentage of participants seroconverting for Anti Nucleoprotein antibodies | Month 6
  (qualitative Elisa)
Percentage of participants seroconverting for Anti Nucleoprotein antibodies | Month 12
  (qualitative Elisa)
Percentage of participants seroconverting for Anti Nucleoprotein antibodies | Month 24
  (qualitative Elisa)
Seroconversion or increase of factor 2 titer of antibodies anti-Spike/anti-RBD between the second and the third dose for the participants with 3 injections | Month 1 after the third dose
  (qualitative Elisa)
Seroconversion or increased levels of anti-Spike/anti-RBD antibodies between the last injection of the initial vaccine regimen and the booster dose | Month 1 after the booster dose
  (qualitative Elisa)

SECONDARY OUTCOMES:
These secondary outcome only concern the adult cohort. Cellular immunity to Covid-19 vaccination | Inclusion
  ELISpot Test
Cellular immunity to Covid-19 vaccination | Month 6
  ELISpot Test
Cellular immunity to Covid-19 vaccination | Month 24
  ELISpot Test
For participants with first injection with Astra-Zeneca vaccine AZD1222 and second injection with Pfizer ARNm vaccine BNT161b2 : humoral and cellular immunity to Covid-19 vaccination | Inclusion
  qualitative Elisa and ELISpot Test
For participants with first injection with Astra-Zeneca vaccine AZD1222 and second injection with Pfizer ARNm vaccine BNT161b2 : humoral and cellular immunity to Covid-19 vaccination | Month 1
  qualitative Elisa and ELISpot Test
For participants with first injection with Astra-Zeneca vaccine AZD1222 and second injection with Pfizer ARNm vaccine BNT161b2 : collection of immediate adverse effects | within 15 minutes after injection of Pfizer ARNm vaccine
  collection by a self-monitoring log
For participants with first injection with Astra-Zeneca vaccine AZD1222 and second injection with Pfizer ARNm vaccine BNT161b2 : collection of adverse effects expected from the database | within 7 days after injection of Pfizer ARNm vaccine
  collection by a self-monitoring log
For participants with first injection with Astra-Zeneca vaccine AZD1222 and second injection with Pfizer ARNm vaccine BNT161b2 : collection of adverse effects | within 28 days after injection of Pfizer ARNm vaccine
  collection by a self-monitoring log

CONTACTS AND LOCATIONS:
Overall Officials: Linda Wittkop, MDPhD, Principal Investigator — CHU de Bordeaux, Université de Bordeaux; Paul Loubet, MDPhD, Principal Investigator — CHU de Nimes, Université de Nimes; Odile Launay, MDPhD, Principal Investigator — Assistance Publique des Hôpitaux de Paris, Université de Paris; Romain Basmaci, MDPhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (3):
- France (3):
  - Cmg-Ec U1219, Bordeaux
  - Nîmes CHU, Nîmes
  - Paris Cochin APHP, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chalouni M, Loubet P, Lhomme E, Ninove L, Barrou B, Blay JY, Hourmant M, de Seze J, Laville M, Laviolle B, Lelievre JD, Morel J, Quoc SN, Spano JP, Terrier B, Thiebaut A, Viallard JF, Vrtovsnik F, Circosta S, Barquin A, Gharib M, Tartour E, Parfait B, Thiebaut R, Meyer L, de Lamballerie X, Launay O, Wittkop L; ANRS0001S COV-POPART study group. Association between humoral serological markers levels and risk of SARS-CoV-2 infection after the primary COVID-19 vaccine course among ANRS0001S COV-POPART cohort participants. BMC Infect Dis. 2024 Sep 27;24(1):1049. doi: 10.1186/s12879-024-09861-5. PMID 39333909
- See also: communication to the general public — https://www.covireivac.fr/vous-allez-etre-vaccine-contre-la-covid-19-faites-progresser-les-connaissances-en-participant-a-la-cohorte-anrs-cov-popart/
- See also: press release — https://www.anrs.fr/fr/presse/communiques-de-presse/801/la-recherche-vaccinale-covid-19-se-poursuit-au-sein-de-la